CLINICAL TRIAL: NCT06450015
Title: Comparison of Vacuum Assisted Closure and Saline Dressing in Patients With Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children Hospital and Institute of Child Health, Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Adeel Ashiq, Principal Investigator, Children Hospital and Institute of Child Health, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: adeel6
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: effectiveness of Vacuum Assisted Closure therapy with saline dressing in management of diabetic foot ulcers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vacuum Assisted Closure therapy (Experimental): Diabetic wounds managed wit VAC dressing
  Interventions: Device: Vacuum Assisted Closure
- Saline Dreesing (Experimental): Saline dressing was done in these patients
  Interventions: Other: Saline Dressing

INTERVENTIONS:
Device: Vacuum Assisted Closure — VAC applied after debridement and saline packing
  Arms: Vacuum Assisted Closure therapy
Other: Saline Dressing — Wound was managed by saline dressing
  Arms: Saline Dreesing

SUMMARY:
Conventionally diabetic foot is treated with moist wound dressing and antibiotics but recent studies show that VAC dressing gives better results as compared to conventional saline dressing in treating Diabetic Foot Ulcers. This may decrease amputations rate, work load on hospitals, hospital stay, repeated hospital admissions, unemployment and can improve patient's quality of life. Objective of the study was to compare the effectiveness of Vacuum Assisted Closure therapy with saline dressing in management of diabetic foot ulcers in terms of granulation tissue formation and wound healing.

DETAILED DESCRIPTION:
it was a randomized Controlled Trial done in department of Surgery, Mayo Hospital,vLahore, Pakistan from January 2022 to July 2022. Patients divided in two groups, in the VAC group (Group A), the wound bed was filled with a saline soaked gauze piece after it is thoroughly cleaned. VAC was applied by placing sterile pads in two layers with a 16Fr Ryle's tube placed between the two layers and then the wound was sealed by a sterile transparent polyurethane sheet. The tube was connected to a wall mounted suction device and the pressure was set at -125 mmHg. In the Saline group (Group B), normal saline dressing was given. This consists of placing a saline soaked gauze piece over the wound bed after cleaning the wound. Patients were assessed and followed for wound healing. The primary outcome parameter was time taken to complete wound healing. Secondary outcome parameters were granulation tissue formation using a visual score and complication of bleeding, pain, and infection. Only healthy granulation tissue which appears pink was considered for scoring assessment. Infection was assessed by wound culture sensitivity which was sent every week.

ELIGIBILITY:
Inclusion Criteria:

* • Diabetic foot ulcer (DFU) patients between the ages of 18 and 60

  * Patients of both genders
  * Diabetic foot ulcer (DFU) patients whose ulcers are smaller than 15 cm in diameter.

Exclusion Criteria:

* • Coagulopathy

  * Venous diseases
  * Foot Ulcers with underlying Osteomyelitis
  * Charcot's joint
  * Peripheral Vascular Diseases
  * Patients with Wegener's Grade IV
  * Involving both feet
  * Patients with HIV and Chronic Liver Disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
time to wound healing | 1 month
  total time for wound healing was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Ashiq, MS, Principal Investigator — The Children Hospital
Locations (1):
- The Children Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Not sharing